CLINICAL TRIAL: NCT02612961
Title: Normal Saline Use With Suctioning: A Randomized-Controlled Trial - Pilot Study
Brief Title: Normal Saline Use With Suctioning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00054395
Record Dates: First submitted 2015-11-18; First posted 2015-11-24 (Estimated); Last update posted 2018-02-26 (Actual); Status verified 2018-02

CONDITIONS: Tracheostomy
Keywords: Mechanically ventilated patients; Normal Saline; Tracheostomy Tube Suctioning
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Saline Instillation (Experimental): 3mL normal saline from pink sodium chloride bullet instilled into tracheostomy immediately prior to suctioning.
  Interventions: Other: 3mL of normal saline from the pink sodium chloride bullet
- Placebo (Sham Comparator): Pretend to instill 3mL of normal saline using empty pink sodium chloride bullet immediately prior to suctioning.
  Interventions: Other: Sham Comparator of 3mL normal saline

INTERVENTIONS:
Other: 3mL of normal saline from the pink sodium chloride bullet
  Arms: Saline Instillation
Other: Sham Comparator of 3mL normal saline
  Arms: Placebo

SUMMARY:
A long-standing intervention during tracheostomy tube suctioning in acute care settings is use of saline to loosen and remove respiratory tract secretions, maintain airway patency, and prevent mucus plugs. Controversy exists regarding safely using saline prior to suctioning for head and neck cancer and mechanically ventilated patients. To date, all studies had methodological limitations. In 2013, the clinical consensus statement published by AAO-HNSF identified a research gap based on lack of strong scientific evidence. A single site, randomized controlled pilot study will be conducted to evaluate effects of saline instillation with tracheostomy tube suctioning; test feasibility of proposed methods and procedures; and ensure proposed outcome variables are measurable and not confounded by extraneous variables. Institutional review board approval will be obtained before eligible adult subjects (inpatient and intensive care units) are recruited and consented. Oxygen saturation and heart rate are primary outcome variables; secondary outcome variables are mucus plugs and ventilator-associated pneumonias; other demographic data and patient characteristic variables; and outcome variables on complications and length of stay. Mean, standard deviation, median, and interquartile range will be calculated for continuous variables using t-tests to compare pre- and post-assessment scores. Frequencies and percentages will be calculated for categorical variables using Chi square and Fisher Exact tests to compare pre- and post-assessment scores. Multiple regression analysis will be used to control for confounding variables. This study is innovative as the first to recruit both head and neck cancer patients and mechanically ventilated patients and to measure all major outcomes of interest in one study. Understanding the effects of normal saline instillation will enable development of evidence-based guidelines and standardized protocols for tracheostomy tube suctioning.

ELIGIBILITY:
Inclusion Criteria:

* Adult Patients, ages 18 or older, cared for on adult inpatient units/wards.
* Patients who have a tracheostomy tube.
* Tracheostomy tube has been in place at lease for 72 hours (to avoid any late effects of anesthesia that was administered at the time of tracheostomy tube placement).
* Patients must have a physician order to suction the tracheostomy tube at least every 8 hours. This will help us to recruit patients for whom suctioning is already part of standard care. Therefore, patients will not undergo unnecessary suctioning for the purpose of the study.
* Expected hospitalization to be 5 days or greater after consent.

Exclusion Criteria:

* Fresh tracheostomy that still has bleeding from the stoma (< 72 hours since the surgical placement of a tracheostomy tube).
* Active respiratory distress or hemodynamic changes that warrant a change in the existing treatment plan.
* Patients who are expected to die or undergo withdrawal of treatment within 48 hours.
* Patients who are allergic to latex to avoid a reaction with the red rubber suction catheter that will be used in the study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-01-16 (Actual); Study Completion 2016-01-16 (Actual)

PRIMARY OUTCOMES:
Change in Oxygen Saturation | immediately prior to intervention, immediately after intervention, immediately after suctioning patient, again at 1-minute and 5-minute post-suction. Repeated 3 times daily for 5 consecutive days
Change in Heart Rate | immediately prior to intervention, immediately after intervention, immediately after suctioning patient, again at 1-minute and 5-minute post-suction. Repeated 3 times daily for 5 consecutive days

SECONDARY OUTCOMES:
Quality of Life Questionnaire for Mechanically Ventilated ICU patients | 5 Days
  12 item questionnaire developed for patients who are mechanically ventilated or patients with a tracheostomy tube who are not mechanically ventilated.
Patient's Experience with Normal Saline Instillation and Tracheostomy Tube Suctioning Questionnaire. | 5 Days
  5 item questionnaire developed to assess patient's experience with normal saline instillation.
Change in Blood Pressure | immediately prior to intervention, immediately after suctioning patient, again at 1-minute and 5-minute post-suction. Repeated 3 times daily for 5 consecutive days
  Systolic and Diastolic Blood pressure
Secretion Volume measured after suctioning patient. | 5 days

OTHER OUTCOMES:
Assessment for Presence of Mucus Plug in tracheostomy tube lumen. | 5 Days
  visual assessment of tracheostomy tube for presence of mucus plug.
Length of stay in the intensive care unit, wards, hospital. | through study completion, an average of 1 year.
  identified by assessing patient's electronic health record.
Presence of Ventilator Associated Pneumonia based on Center for Disease Control algorithm for clinically defined pneumonia. | through study completion, an average of 1 year
  Identified based on presence of new infiltrates on chest X-rays, fever > 38°F, Leukopenia (<4000 WBC/mm-squared), or Leukocytosis (≥12,000WBC/mm-squared), positive sputum cultures, and worsening gas exchange documented in patient's electronic health record based on the Center for Disease Control algorithm for clinically defined pneumonia.
Time Duration of mechanical ventilation identified through patient's electronic health record. | through study completion, an average of 1 year.
Patient presentation of Dyspnea with saline instillation, assessed by patient's presentation, visual assessment. | 5 Days
change in presence of bleeding through tracheostomy tube during intervention, assessed visually. | prior to saline instillation and post suctioning of patient, 3 times daily for 5 consecutive days.
Presence of atelectasis in patient assessed via Chest X-ray in patient's electronic record. | 5 days
presence of tracheitis in patient assessed from patient's electronic record. | 5 days

CONTACTS AND LOCATIONS:
Locations (1):
- The Johns Hopkins Hospital, Baltimore, Maryland, United States

REFERENCES:
- [Background] Halm MA, Krisko-Hagel K. Instilling normal saline with suctioning: beneficial technique or potentially harmful sacred cow? Am J Crit Care. 2008 Sep;17(5):469-72. No abstract available. PMID 18776003
- [Background] Paratz JD, Stockton KA. Efficacy and safety of normal saline instillation: a systematic review. Physiotherapy. 2009 Dec;95(4):241-50. doi: 10.1016/j.physio.2009.06.002. Epub 2009 Sep 12. PMID 19892088
- [Background] Dennis-Rouse MD, Davidson JE. An evidence-based evaluation of tracheostomy care practices. Crit Care Nurs Q. 2008 Apr-Jun;31(2):150-60. doi: 10.1097/01.CNQ.0000314475.56754.08. PMID 18360145
- [Background] American Association for Respiratory Care. AARC Clinical Practice Guidelines. Endotracheal suctioning of mechanically ventilated patients with artificial airways 2010. Respir Care. 2010 Jun;55(6):758-64. PMID 20507660
- [Background] Mitchell RB, Hussey HM, Setzen G, Jacobs IN, Nussenbaum B, Dawson C, Brown CA 3rd, Brandt C, Deakins K, Hartnick C, Merati A. Clinical consensus statement: tracheostomy care. Otolaryngol Head Neck Surg. 2013 Jan;148(1):6-20. doi: 10.1177/0194599812460376. Epub 2012 Sep 18. PMID 22990518
- [Background] Caruso P, Denari S, Ruiz SA, Demarzo SE, Deheinzelin D. Saline instillation before tracheal suctioning decreases the incidence of ventilator-associated pneumonia. Crit Care Med. 2009 Jan;37(1):32-8. doi: 10.1097/CCM.0b013e3181930026. PMID 19050607
- [Background] Reeve JC. Instillation of normal saline before suctioning reduces the incidence of pneumonia in intubated and ventilated adults. Aust J Physiother. 2009;55(2):136. doi: 10.1016/s0004-9514(09)70044-3. PMID 19534012
- [Background] Kleinpell R. Use of Normal Saline Instillation with Suctioning: The Debate Continues. Critical Care Alert 2009;17(1):1.
- [Background] Christensen RD, Henry E, Baer VL, Hoang N, Snow GL, Rigby G, Burnett J, Wiedmeier SE, Faix RG, Eggert LD. A low-sodium solution for airway care: results of a multicenter trial. Respir Care. 2010 Dec;55(12):1680-5. PMID 21122176
- [Background] Maggiore SM, Lellouche F, Pignataro C, Girou E, Maitre B, Richard JC, Lemaire F, Brun-Buisson C, Brochard L. Decreasing the adverse effects of endotracheal suctioning during mechanical ventilation by changing practice. Respir Care. 2013 Oct;58(10):1588-97. doi: 10.4187/respcare.02265. Epub 2013 Mar 6. PMID 23466423
- [Background] Evans J, Syddall S, Butt W, Kinney S. Comparison of open and closed suction on safety, efficacy and nursing time in a paediatric intensive care unit. Aust Crit Care. 2014 May;27(2):70-4; quiz 75-6. doi: 10.1016/j.aucc.2014.01.003. Epub 2014 Mar 11. PMID 24636425
- [Background] Iranmanesh, Sedigheh, Rafiei, Hossein. Normal saline instillation with suctioning and its effect on oxygen saturation, heart rate, and cardiac rhythm. Int J Nurs Educ 2011;3(1):42.
- [Background] Caparros AC. Mechanical ventilation and the role of saline instillation in suctioning adult intensive care unit patients: an evidence-based practice review. Dimens Crit Care Nurs. 2014 Jul-Aug;33(4):246-53. doi: 10.1097/DCC.0000000000000049. PMID 24895955